CLINICAL TRIAL: NCT00547612
Title: Pilot Trial of the NK1 Receptor Radio-Ligand [18F]SPA-RQ: Imaging Pancreatic Ductal Adenocarcinoma
Brief Title: Positron Emission Tomography Using [18F]-Labeled Substance P Antagonist Receptor Quantifier in Finding Disease in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Diagnostic
Other Study IDs: 070222; 07-C-0222; CDR0000570181
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chromatography, High Pressure Liquid

INTERVENTIONS:
Other: high performance liquid chromatography
Other: pharmacological study
Radiation: [18F]-labeled substance P antagonist receptor quantifier

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET) using [18F]-labeled substance P antagonist receptor quantifier, may be effective in finding disease in patients with pancreatic cancer.

PURPOSE: This phase I trial is studying how well a PET scan using [18F]-labeled substance P antagonist receptor quantifier works in finding disease in patients with pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether [18F]-labeled substance P antagonist receptor quantifier positron emission tomography can identify pancreatic cancer evident on multiphase CT scan.

OUTLINE: Patients undergo multiphase CT scan of the chest, abdomen, and pelvis. No more than 15 days later, patients receive [18F]-labeled substance P antagonist receptor quantifier IV and undergo positron emission tomography over 6 hours.

Blood is collected periodically to measure the metabolism of the radiotracer by high performance liquid chromatography with radioactive detectors.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Primary or metastatic disease
* At least one site of measurable disease
* Enrolled in an NCI protocol (either a treatment or screening protocol) such as NCI-05-C-0044 or NCI-05-C-0141

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* WBC ≥ 1,200/mm³
* Creatinine < 2.0 mg/dL
* Negative pregnancy test
* Fertile patients must agree to use effective contraception
* Not pregnant or nursing

Exclusion criteria:

* Allergy to IV contrast
* Claustrophobia that would preclude completion of a scan or unable to lie on one's back for positron emission tomography scan

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* More than 4 weeks since prior abdominal surgery

Exclusion criteria:

* Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits
* Aprepitant within 72 hours of [18F]-labeled substance P antagonist receptor quantifier positron emission tomography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of tumors detected by [18F]-labeled substance P antagonist receptor quantifier positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Royal, MD, FACS, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States